CLINICAL TRIAL: NCT02630095
Title: Effect of Anticoagulation After Endoscopic Therapy in Cirrhotic Patients With Portal Vein Thrombosis：A Zelen-design Multicenter Randomized Controlled Trial
Brief Title: The Effect of Anticoagulation in Cirrhotic Patients With Portal Vein Thrombosis：A Multicenter RCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Public Health Clinical Center (Other Government); ShuGuang Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Pudong New Area Gongli Hospital (Other); Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, Director of department of Gastroenterology, Zhongshan Hospital, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSY-LSX02-2015
Record Dates: First submitted 2015-12-08; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Portal Vein Thrombosis; Liver Cirrhosis
Keywords: anticoagulation
MeSH Terms: conditions — Liver Cirrhosis | interventions — Nadroparin; Warfarin; Ultrasonography, Doppler

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control. (Other): No anticoagulation，just routine follow up.
  Interventions: Device: Doppler ultrasound and CT
- Anticoagulation (Experimental): Nadroparin Calcium and Warfarin
  Interventions: Drug: Nadroparin Calcium and Warfarin; Device: Doppler ultrasound and CT

INTERVENTIONS:
Drug: Nadroparin Calcium and Warfarin — Patients will take warfarin started at a dose of 2.5mg/d and with titration of dose to maintain a target INR of 2-3, and during the of perioperative period of Endoscopic treatment changing to use Nadroparin Calcium 4100IU／d，subcutaneous.
  Arms: Anticoagulation
Device: Doppler ultrasound and CT — all patient will take Doppler ultrasound examination every 3 months ；Abdominal CT will be done every 6 months。

SUMMARY:
The purpose of this study is to determine the effect and safety of anticoagulation after endoscopic therapy in cirrhotic patients with portal vein thrombosis and to explore its effect on long-term rebleeding rate and mortality.

DETAILED DESCRIPTION:
The treatment of cirrhotic patients with PVT (portal vein thrombosis) is clearly recommended in guideline now. Several published studies has confirm the effect and safety of anticoagulation therapy in cirrhotic patients with PVT.The present studies are most observation studies with small sample size and low quality. The investigators need more high-quality research such as randomized controlled trials. This is a Zelen-designed multicenter randomized controlled trial. Patients will randomly enter into two groups:the anticoagulation group or the control group and then the investigator will make sure wether their are fond of the group and make decision by themselves. The recanalization rate and complications will be analyzed

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years old;
* A clinical, radiological or histologic diagnosis of Liver cirrhosis and portal hypertension;
* Diagnosed of Portal vein thrombosis;
* Capable of understanding the purpose and risks of the study and informed consent to participate in the study;
* Have undergone endoscopy to prevent variceal rebleeding.

Exclusion Criteria:

* Age <18 or >70 years;
* Portal vein thrombosis diagnosed before 6 months;
* Patients with signs of acute PVT such as fever，abdominal pain or intestinal obstruction，who should be treated immediately;
* Pregnant or nursing;
* Hepatocellular carcinoma or other cancer;
* Severe cardiopulmonary diseases or concomitant renal insufficiency;
* cavernous transformation of the portal vein;
* Contradictions to endoscopy;
* Contradictions to anticoagulation,such as:allergy to LMWH or warfarin, severe uncontrolled hypertension, history of hemorrhagic cerebral vascular accident, recent peptic ulcer disease, bacterial endocarditis, ulcerative colitis，sustained platelet count < 50 x10^9/L);
* Taking immunosuppressive agent;
* Coagulation disorders other than the liver disease related;
* Variceal bleeding failed to control.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Recanalization rate of PVT | through study completion，an average of 18 months
  Patients will receive Doppler ultrasound and CT before enrolled and followed up by Doppler ultrasound every 3 months ,by CT every 6 months after enrolled，untill the end of the study.

SECONDARY OUTCOMES:
Rebleeding rate | through study completion，an average of 18 months
  The investigators observe the variceal rebleeding events during the study
Incidence rate of complications | through study completion，an average of 18 months
  The investigators observe any severe adverse events caused by anticoagulation therapy or the progress of thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, Professor, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China